CLINICAL TRIAL: NCT04238936
Title: Levels of New Inflammatory Markers in GDM Patients; Serum Amyloid A and Interleukin-1 (IL-1) Receptor Antagonist
Brief Title: GDM Patients and Serum Amyloid A and Interleukin-1 (IL-1) Receptor Antagonist
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, Pınar kadirogullari, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK-2020/02
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Serum amyloid A; Interleukin-1 (IL-1) receptor antagonist
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group ; Patients with gestational diabetes: Women who are diagnosed with GDM between the ages of 18 and 43 will receive blood in the biochemistry tube. This tube will then be centrifuged. A-SAA and IL-1Ra levels will be checked by ELISA method in serum stored at -80 degrees.
  Interventions: Diagnostic Test: Serum amyloid A values; Diagnostic Test: Interleukin-1 (IL-1) receptor antagonist values (A-SAA and IL-1Ra)
- control group ; healthy pregnant women: Women who are healthy pregnant women, the ages of 18 and 43 will receive blood in the biochemistry tube. This tube will then be centrifuged. A-SAA and IL-1Ra levels will be checked by ELISA method in serum stored at -80 degrees.
  Interventions: Diagnostic Test: Serum amyloid A values

INTERVENTIONS:
Diagnostic Test: Serum amyloid A values — Women who are diagnosed with GDM between the ages of 18 and 43 will receive blood in the biochemistry tube. This tube will then be centrifuged. A-SAA and IL-1Ra levels will be checked by ELISA method in serum stored at -80 degrees.
Diagnostic Test: Interleukin-1 (IL-1) receptor antagonist values (A-SAA and IL-1Ra) — Women who are diagnosed with GDM between the ages of 18 and 43 will receive blood in the biochemistry tube. This tube will then be centrifuged. A-SAA and IL-1Ra levels will be checked by ELISA method in serum stored at -80 degrees.
  Groups: study group ; Patients with gestational diabetes

SUMMARY:
Serum amyloid A and Interleukin-1 (IL-1) receptor antagonist (A-SAA and IL-1Ra) values;

* Comparison of pregnant women with and without GDM diagnosis
* Comparison of insulin therapy and diet-regulated GDM patients
* Comparison of pregnant women with and without LGA (large gestational age)
* Comparison of pregnant women with and without polyhydroamnios
* Investigation of its effect on pregnancy prognosis
* In the prediction of GDM diagnosis, it is aimed to study the sensitivity and specificity of both parameters and cut off values.

(In GDM patients, liver and kidney function parameters will also be evaluated with A-SAA and IL-1Ra levels).

ELIGIBILITY:
Inclusion Criteria:

* Patients with 50 gr OGTT + 100 gr OGTT + at 24-28 weeks of gestation
* Patients with 75 gr OGTT + at 24-28 weeks of gestation
* 18-42 years pregnant women

Exclusion Criteria:

* any infection
* Any known fetal chromosomal or structural anomaly
* Preterm membrane rupture
* Preterm delivery
* Preeclampsia or eclampsia
* Placenta previa

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Serum amyloid A (SAA) and Interleukin-1 (IL-1) receptor antagonist level will be examined in the study group consisting of pregnant women with GDM diagnosis and in the control group consisting of healthy pregnant women.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Serum amyloid A | 1 week
  Its level will be checked in the study group consisting of pregnant women with GDM and in the control group consisting of healthy pregnant women.
Interleukin-1 (IL-1) receptor antagonist | 1 week
  Its level will be checked in the study group consisting of pregnant women with GDM and in the control group consisting of healthy pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)